CLINICAL TRIAL: NCT02954432
Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Transcranial Ultrasound (TUS) on the Perception of Pain and Functional Limitations Due to Non-Specific Chronic Low Back Pain (NSCLBP).
Brief Title: Effects of tDCS and TUS on the Perception of Pain and Functional Limitations Due to Non-Specific Chronic Low Back Pain
Status: Active, not recruiting | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P001956
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Chronic Low Back Pain
Keywords: transcranial Direct Current Stimulation; Transcranial Ultrasound; non-invasive brain stimulation
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Phase II
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Active tDCS + Active TUS (Experimental): Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Transcranial Ultrasound (TUS)
- Sham tDCS + Sham TUS (Sham Comparator): Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Transcranial Ultrasound (TUS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — Subjects will receive 20 minutes of either active or sham tDCS at an intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
Device: Transcranial Ultrasound (TUS) — Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.

SUMMARY:
The purpose of this study is to assess the effects of tDCS in combination with TUS for the treatment of pain and functional limitations in subjects with NSCLBP. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study
2. Subjects between 18 to 85 years old
3. Subjects having non-specific chronic low back pain with existing pain for at least 3 months and having pain on at least half the days in the past 6 months with an average of at least 3 on a 0-10 visual analog scale (VAS) scale
4. Pain resistant (partial or no response) to common analgesics and medications for chronic pain used as initial pain management such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, and Codeine.
5. Must have the ability to feel sensation by Von-Frey fiber on the forearm

Exclusion Criteria:

1. Subject is pregnant
2. Contraindications to tDCS in conjunction with TUS, i.e. metallic implant in the brain or implanted brain medical devices
3. History of alcohol or drug abuse within the past 6 months as self reported
4. Use of carbamazepine within the past 6 months as self reported
5. Suffering from severe depression (with a score of >30 in the Beck Depression Inventory)
6. History of neurological disorders as self reported
7. History of unexplained fainting spells as self reported
8. History of severe head injury resulting in more than a momentary loss of consciousness as self reported
9. History of neurosurgery as self reported
10. Unstable pain
11. Large placebo responder
12. Low adherence during the run-in period
13. Low baseline pain

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Teixeira PEP, Pacheco-Barrios K, Uygur-Kucukseymen E, Machado RM, Balbuena-Pareja A, Giannoni-Luza S, Luna-Cuadros MA, Cardenas-Rojas A, Gonzalez-Mego P, Mejia-Pando PF, Wagner T, Dipietro L, Fregni F. Electroencephalography Signatures for Conditioned Pain Modulation and Pain Perception in Nonspecific Chronic Low Back Pain-An Exploratory Study. Pain Med. 2022 Mar 2;23(3):558-570. doi: 10.1093/pm/pnab293. PMID 34633449

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 subjects were enrolled and randomized
Groups:
- Active tDCS + Active TUS: Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
- Sham tDCS + Sham TUS: Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2 milliamps (mA0. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
Period: Overall Study
Arm/Group | Active tDCS + Active TUS | Sham tDCS + Sham TUS
Started | 20 | 20
Completed | 12 | 11
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Population: Baseline for randomized subjects (phase II)
Groups:
- Active tDCS + Active TUS - Phase II: Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
- Sham tDCS + Sham TUS - Phase II: Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
- Total: Total of all reporting groups
Arm/Group | Active tDCS + Active TUS - Phase II | Sham tDCS + Sham TUS - Phase II | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (18.6) | 47.3 (15.7) | 48.2 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: one subject did not declare sex
  Participants
    number analyzed (Participants) | 20 | 19 | 39
    Female | 6 | 14 | 20
    Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 13 | 13 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mechanical Temporal Summation (Hand)
Description: Changes in Mechanical Temporal Summation (TS) from hand will be measured in order to determine whether anodal transcranial direct current stimulation (tDCS) in conjunction with transcranial ultrasound (TUS) is effective in reducing pain of subjects with non-specific chronic low back pain.
Time Frame: Baseline and 3.5 months
Measure: Mean (Standard Error); unit: TSPS percentage change
Groups:
- Sham tDCS + Sham TUS: Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
Arm/Group | Active tDCS + Active TUS | Sham tDCS + Sham TUS
Number analyzed (Participants) | 20 | 20
TSPS percentage change | 15 (8) | -4 (9)

2. Primary Outcome: Changes in Conditional Pain Modulation (Hand)
Description: Changes in Conditional Pain Modulation (CPM) will be measured in the hand in order to determine whether anodal transcranial direct current stimulation (tDCS) in conjunction with transcranial ultrasound (TUS) is effective in increasing the pain pressure threshold in subjects with non-specific chronic low back pain.
Time Frame: Baseline and 3.5 months
Measure: Mean (Standard Error); unit: CPM percentage changes
Arm/Group | Active tDCS + Active TUS | Sham tDCS + Sham TUS
Number analyzed (Participants) | 20 | 20
CPM percentage changes | 94 (22) | -4 (19)

3. Primary Outcome: Changes in Pain
Description: Changes in the Visual Analogue Scale (VAS) for pain will be measured in order to measure any changes in pain levels when subjects come in for sessions.
Time Frame: Baseline and 3.5 months
Measure: Mean (Standard Error); unit: percentage changes
Arm/Group | Active tDCS + Active TUS | Sham tDCS + Sham TUS
Number analyzed (Participants) | 20 | 20
percentage changes | 45 (2.4) | 24 (2)

ADVERSE EVENTS:
Time Frame: 3.5 months
Description: Adverse effects were collected with a questionnaire for adverse effects
Groups:
- Active tDCS + Active TUS: Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of active tDCS at intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of active TUS. During active stimulation the ultrasound will be active for the full 20 minutes.
- Sham tDCS + Sham TUS: Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  transcranial Direct Current Stimulation (tDCS): Subjects will receive 20 minutes of sham tDCS at intensity of 2 milliamps (mA). The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Transcranial Ultrasound (TUS): Subjects will receive 20 minutes of sham TUS. During sham stimulation the ultrasound will not be active for the full 20 minutes.
Arm/Group | Active tDCS + Active TUS | Sham tDCS + Sham TUS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 15/20 | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS + Active TUS (N=20) | Sham tDCS + Sham TUS (N=20)
tingling (Nervous system disorders) | 15 (102) | 13 (74) — tingling at the site of stimulation event (mild)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT02954432/Prot_SAP_000.pdf